CLINICAL TRIAL: NCT04726566
Title: Return to Sport and Functional Assessment After Surgery for Chronic Lateral Ankle Instability
Brief Title: Chronic Ankle Instability Return to Sport
Acronym: CAIRTS
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-A00154-35
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Ankle Instability
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroscopic stabilization: Patient will have an anatomical surgery of chronic lateral ankle instability under arthroscopy
  Interventions: Procedure: Tendon graft; Procedure: Suture with biological reinforcement

INTERVENTIONS:
Procedure: Tendon graft — Anatomical surgery for chronic lateral ankle instability under arthroscopy with tendon graft
Procedure: Suture with biological reinforcement — Anatomical surgery for chronic lateral ankle instability under arthroscopy by suture with biological reinforcement

SUMMARY:
Real-life, observational, monocentric, prospective, longitudinal study, carried out at the European Center for Sports Rehabilitation (CERS), France.

DETAILED DESCRIPTION:
The data will be collected through an electronic Case Report Form completed by the physician, and some auto-questionnaire completed by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 15 years;
* Patient treated at the European Sports Rehabilitation Center after a first arthroscopic surgery on the external lateral ligament of the ankle for chronic instability by anatomical reconstruction:

  * With tendon graft;
  * By suture with biological reinforcement;
* Non-opposition of the patient and his/her parents (if minor) to the collection of his/her personal data.

Exclusion Criteria:

- Minor patient (age <18 years) not accompanied by one of his/her parents or legal representative during the inclusion visit;

* History of surgery on the same ankle;
* Associated complex osteochondral or internal ligament damage, syndesmosis, fracture;
* Non-anatomical reconstruction;
* Inability of the patient to understand the study protocol;
* Vulnerable person whose inclusion is not justified by the purposes of the research: pregnant woman, person undergoing psychiatric care, or adult person subject to legal protection.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in rehabilitation at the European Sports Rehabilitation Center after anatomical surgery for chronic lateral ankle instability.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Rate of return to main sport at the expected level in both groups | 10 months
  The main objective is to evaluate the rate of patients who returned to sport at the level before the injury, according to their evaluation, 10 months after arthroscopic stabilization according to the surgical technique used (repair by suture or reconstruction by tendon graft).

SECONDARY OUTCOMES:
Factors associated with the lack of resumption of sport at the level before the injury | 10 months
  Factors associated with the lack of resumption of sport at 10 months at the level before the injury
Time taken to resume sport after arthroscopic stabilization | 10 months
  Evaluate the time taken to resume sport after arthroscopic stabilization according to the surgical technique used
Functional state of the ankle | 10 months
  Evaluate the functional state of the ankle and the level of activity of the patients during the follow-up according to the surgical technique used

CONTACTS AND LOCATIONS:
Locations (1):
- European sports rehabilitation center, Capbreton, France

IPD SHARING:
Plan to Share IPD: No